CLINICAL TRIAL: NCT01031303
Title: Immunogenicity and Safety of the Sanofi Pasteur's DTacP-IPV Combined Vaccine (TETRAXIM™) Given as a Booster Dose at 4 to 6 Years of Life in Children Previously Vaccinated With PENTAXIM™ in the Study E2I34
Brief Title: Immunogenicity and Safety of TETRAXIM™ Given as a Booster Dose at 4 to 6 Years of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E2I57; UTN: U1111-1112-2680 (Other: WHO)
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis
Keywords: Diphtheria; Tetanus; Pertussis; Poliomyelitis; PENTAXIM™; TETRAXIM™
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Biological: DTacP-IPV combined vaccine (TETRAXIM™)

INTERVENTIONS:
Biological: DTacP-IPV combined vaccine (TETRAXIM™) — 0.5 mL, Intramuscular
  Other Names: TETRAXIM™

SUMMARY:
The purpose of this study is to provide further immunogenicity and safety information of sanofi pasteur's DTacP-IPV combined vaccine (TETRAXIM™) as a booster dose during the 4th and 6th year of life in children that previously received in Study E2I34 (NCT 00255021), sanofi pasteur DTacP-IPV// PRP~T vaccine (PENTAXIM™) as a three-dose primary and booster vaccinations.

Primary Objective :

* To assess immunogenicity in terms of seroprotection rates (Diphtheria, Tetanus, Polio types 1, 2 and 3) and seroconversion/vaccine response rates to acellular Pertussis antigens (Pertussis toxoid [PT], Filamentous Haemagglutinin [FHA]) of sanofi pasteur's DTacP-IPV (Tetraxim™) vaccine, one month after the booster dose given at 4 to 6 years of age.

Secondary Objectives :

* To describe the antibody persistence in terms of anti-pertussis antibody levels (anti-PT, and -FHA) and in terms of seroprotection rates and GMTs for Diphtheria, Tetanus, and Poliovirus types 1, 2 and 3, just before administration of the booster dose (at Visit 1) in all subjects at 4-6 years of age.
* To assess immunogenicity in terms of seroprotection rates (Diphtheria, Tetanus, Polio types 1, 2 and 3) and seroconversion/ vaccine response rates to acellular Pertussis antigens (PT, FHA) of sanofi pasteur's DTacP-IPV (Tetraxim™) vaccine, one month after administration of the booster dose given at 4 to 6 years of age.
* To describe the safety after the booster dose of the study vaccine.

DETAILED DESCRIPTION:
All participants that previously completed the three-dose primary and the booster vaccinations in the study E2I34 (NCT 00255021) will be contacted to enroll in this study to receive sanofi pasteur's DTacP IPV combined vaccine (Tetraxim™) at 4 to 6 years of age.

Participants will receive the study vaccine [sanofi pasteur's DTacP-IPV vaccine (TETRAXIM™)] at 4 to 6 years of age (at visit 1).

ELIGIBILITY:
Inclusion Criteria :

* Aged 4-6 years inclusive on the day of inclusion
* Child having completed the three-dose vaccination and the booster vaccination with DTacP-IPV//PRP~T combined vaccine (PENTAXIM™) of the study E2I34
* Informed consent form signed by the parent(s) or other legal representative
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria :

* Participation in another clinical trial in the 4 weeks preceding the trial inclusion
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received in the past or current or planned administration during the trial (including immunoglobulins)
* Any vaccination in the 4 weeks preceding the trial vaccination
* History of diphtheria, tetanus, pertussis, poliomyelitis infection (confirmed either clinically, serologically or microbiologically)
* Clinical or known serological evidence of systemic illness including Hepatitis B, Hepatitis C and/or Human immunodeficiency virus (HIV) infection
* Previous vaccination against the diphtheria, tetanus, pertussis, poliomyelitis diseases infection with the trial vaccine or another vaccine after completion of previous study E2I34
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of/current major neurological diseases or seizures
* Febrile illness (temperature ≥ 38°C) or acute illness on the day of inclusion.
* Serious or severe reaction after a previous dose of any vaccine containing pertussis antigen, such as
* encephalopathy (with or without convulsions) in the 7days following previous administration of a pertussis containing vaccine,
* temperature more than 39.5°C within 48 hours following vaccine injection, not due to another identifiable cause
* inconsolable crying equal or more than 3 hours within 48 hours following vaccine injection,
* hypotonic hyporesponsive episode within 48 hours following vaccine injection,
* seizures with or without fever within 3 days following vaccine injection.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of TETRAXIM™ after booster vaccination. | 30 days post-vaccination

SECONDARY OUTCOMES:
To provide information concerning the safety after booster administration of TETRAXIM™. | 30 days post-vaccination and entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — sanofi pasteur SA
Locations (1):
- Bangkok, Thailand

REFERENCES:
- [Derived] Pancharoen C, Chotpitayasunondh T, Chuenkitmongkol S, Ortiz E. Long-term immunogenicity assessment of a DTaP-IPV//PRP-T vaccine given at 2, 4, 6 and 18-19 months of age, and immunogenicity and safety of a DTaP-IPV vaccine given as a booster dose at 4 to 6 years of age in Thai children. Southeast Asian J Trop Med Public Health. 2012 May;43(3):687-98. PMID 23077849
- See also: Related Info — http://www.sanofipasteur.com